CLINICAL TRIAL: NCT06580600
Title: A Single Centre Randomised, Feasibility Study Using Point-of-care (POC) Testing for Respiratory Viruses to Direct Oral Corticosteroids Use in Preschool-aged Children With Acute Wheeze.
Brief Title: PREcision Medicine Directed Corticosteroids In Children With preSchool Wheeze
Acronym: PRECISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Asthma UK (Other); Pediatric Emergency Research in the UK and Ireland (PERUKI) (Other)
Responsible Party: Principal Investigator, Thomas Waterfield, Clinical Lecturer in Paediatrics, Queen's University, Belfast
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B24/01
Record Dates: First submitted 2024-08-07; First posted 2024-08-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Wheezing
Keywords: pre-school; wheeze; corticosteroid; point-of-care
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Intervention Model Description: randomised (1:1) to receive OCS or No OCS (both of which are standard of care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCS (Active Comparator): To receive OCS (this is standard of care as the children will be recruited if their is clinicial uncertainty over the benefit of OCS, i.e. this is not a CTIMP). The local policy is to prescribe Dexamethasone suspension 300mcg/kg in a single dose.
  Interventions: Diagnostic Test: Point of care respiratory virus testing
- No OCS (No Intervention): The child will not recieve any cortisteroid medications (this is standard of care as the children will be recruited if their is clinicial uncertainty over the benefit of OCS, i.e. this is not a CTIMP).

INTERVENTIONS:
Diagnostic Test: Point of care respiratory virus testing — Patients to be randomised to receive OCS based on the the result of the RSV results within their respiratory virus test. This test will be performed as a point of care (POC) test in ED.
  This intervention will stratify the randomisation in a 1:1 ratio, to receive OCS or not.
  NB) Whilst the respiratory pathogen test is not routine care to determine the OCS prescription, it is frequently used within this setting. Additionally both the receipt (or not the receipt) of OCS is within standard care pathway. For the purpose of the trial OCS = Dexamethasone, which is delivered as oral suspension 300mcg/kg as per standard practice within the local Trust.
  Other Names: RSV test
  Arms: OCS

SUMMARY:
Young children frequently attend the emergency department (ED) with wheeze which is usually triggered by a virus infection, such as the common cold. Wheeze can be treated with inhaled medications and sometimes oral steroid medicines are also given to reduce swelling within the lungs. Unfortunately, oral steroids can have side effects. Despite lots of research there is no clear evidence that oral steroids work in young children with a wheeze attack. It is likely that some children get better quicker with oral steroids but deciding who to treat is difficult. This results in differences in care with some children receiving unnecessary oral steroids and others not receiving them when they could benefit.

The investigators hypothesise that in a subgroup of children with mild-to-moderate acute wheeze attacks, the viral trigger can predict their response to steroid medications. Previously, respiratory virus testing was too slow to be used to inform treatments in the ED. Now, point-of-care (POC) viral tests can provide results within 30 minutes. There is a research gap regarding the role of these tests in determining steroid responsiveness and outcomes in children presenting with acute wheeze in the pre-school population.

In order to address the hypothesis in a future definitive trial, the feasibility of using (POC) viral tests to randomise steroid treatments for children in a clinical study in the ED setting must be ascertained. The PRECISE Study will therefore be a single centre randomised, feasibility study enrolling approximately 60 pre-school aged children to inform a future definitive multi-centre Randomised Controlled Trial.

DETAILED DESCRIPTION:
PRECISE will be a feasibility study; conducted as a single-centre, prospective, randomised open-label study. Participants will be screened by the clinical team from attendances to the local Emergency Department (ED). Participants meeting the study inclusion criteria, by age and symptoms, will be entered into a screening log. If the participant is not recruited the reason will be recorded. Participants will be assessed using the inclusion and exclusion criteria (described in other sections). Eligibility will be flagged by a member of the clinical team and then subsequently confirmed by a member of the research team. However, the medical care given to, and medical decisions made on behalf of, participants will be the responsibility of an appropriately qualified treating physician.

The research team member will discuss each eligible participant with their treating physician, to confirm agreement with study enrolment. Parents of eligible children will then be introduced to the research team to provide study information, confirm eligibility, and obtain informed consent. Families will be given time to read the Participant Information Sheets (PIS) and reflect on their discussion with the researcher who will then offer the opportunity to answer further questions. With written informed consent obtained, the participant will be enrolled. This will require the first nasal/nasopharyngeal swab (NPS) to be collected and tested for RSV and other respiratory viral infections. This NPS is for the purposes of the study but results will be made available to the treating clinician and the family. Based on the result of Participants' NPS they will then be randomised to receive oral corticosteroids (OCS) or no OCS through an automated process with a 1:1 ratio. Throughout this process clinicians will continue to perform investigations and administer additional standard of care treatment according to local hospital guidance. Administration of emergency standard of care treatment will not be delayed pending consent discussions or NPS result.

OCS therapy, if given, will be administered as oral dexamethasone according to local standard of care. If the participant vomits within 30 minutes of dexamethasone administration, it may be re-administered at the discretion of the treating clinician. As there is no blinding to the study participants or clinicians regarding the randomisation allocation, the treating clinician may choose to determine the OCS therapy plan at any point after enrolment, irrespective of study randomisation, based on the patient's clinical status.

After the initial ED presentation there are two other time points in the study, i) a review in 2 working days and a phone call at 28 days, post enrolment. UK BTS/SIGN guidance recommends all patients presenting with acute asthma or wheeze should be reviewed following discharge from ED/hospital within two working days. This is not routinely offered locally however, for the purposes of the study, participants will be offered a review with a clinical member of the research team and a repeat nasal swab event will take place. A member of the research team will call parents on day 28 to complete each child's research record.

Additionally, participants may consent to an optional finger prick blood testing at enrolment to elicit their blood eosinophil count using a Point of care (POC) white cell differential device. As with the NPS result, the family and clinicians will be made aware of the result.

Finally parents of participants in the PRECISE study will be invited to take part in semi-structured interviews after the day 28 call for further feasability and acceptability analysis.

ELIGIBILITY:
Inclusion Criteria:

* 24-60 months (infants from 24 months +0 days to 60 months + 0 days inclusive)
* Clinical diagnosis of acute wheeze
* Clinical uncertainty regarding the benefit of OCS as part of patient's standard care

Exclusion Criteria:

* Signs and symptoms of severe or life-threatening wheeze
* Patients presenting with wheeze suspicious for a non - respiratory cause
* Clinical evidence of shock or bacterial sepsis
* Past history of severe or life-threatening asthma or history of previous PICU admission with acute wheeze
* History of preterm birth (before 36+0 weeks gestation)
* Known immunodeficiency/ongoing immunosuppressive therapy
* Contraindication to oral corticosteroids
* Previously enrolled in the PRECISE Study

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Screening Log completed through study completion, (estimated < 1 year)
  Reporting the proportion of eligible patients that are enrolled in the PRECISE Study following screening Reporting all reasons for not screening enrolling any eligible patients.
Adherance | measured at visit 2 and at 28 days post enrolment per patient. Throughout study completion, (estimated < 1 year)
  Reporting the proportion of randomised patients remaining in allocated treatment arm. I.e. how many patients randomised to NOT recieve OCS have received them within 28 days of enrolment.
Timeliness | Timeliness measured on CRFs throughout study completion, (estimated < 1 year)
  The time (minutes) for i) triage to clinician decision regarding eligibility to enrolment ii) screening until availability of POC test results iii) screening to documented time of randomisation iv) screening to documented time of OCS administration (if applicable)
Acceptability | Collected at 2 and 28 days post enrolment per patient. Data collected through study completion, (estimated < 1 year))
  Description of parent/guardian feedback on how acceptable the process of being enrolled and randomised in the study was. This includes a description of perceived barriers to future definitive trial collected from families.

SECONDARY OUTCOMES:
viral aetiology | Through study completion, (estimated < 1 year)
  To describe viral aetiology of preschool wheeze in included cohort. I.e. the proportions of patients with positive respiratory viral tests for RSV and/or other respiratory virus/ or no virus detected. This includes a description of the CT - values associated with positive respiratory viral test results.
Concordance of test results | Between enrolment and the second visit. (Throughout study completion, (estimated < 1 year))
  The proportions of patients with discordant respiratory viral tests over consecutive visits.
Acceptability of tests to formulate plan | Data collected within one month of enrolment. Throughout study completion, (estimated < 1 year)
  To assess parent/guardian acceptability of using a viral POC test in ED to formulate a management plan for pre-school wheeze (using a mixed methods approach).
Acceptability of tests to be repeated in study | Data collected within one month of enrolment. Throughout study completion, (estimated < 1 year)
  To assess the feasibility of obtaining second nasal/nasopharyngeal (NP) swab and achieving follow up at specified time points
Airway immune response | Analysis to be performed within 1 year of study closure.
  Analysis of airway immune responses in preschool wheeze. To describe the immune response associated with preschool wheeeze according to numerous factors, including patient presentation, viral status and OCS use.
blood eosinophil testing in acute setting | measured at enrolment and visit 2 per patient. Analysis to be completed within 6 months of study closure.
  To assess the feasibility of obtaining finger prick blood test for peripheral blood eosinophil - count testing:
  i) proportion of patients taking up optional finger-prick testing ii) describe the peripheral eosinophil count values in patients undergoing optional testing and associations with viral test results and clinical values.

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Groves, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Royal Belfast Hospital for Sick Children, Belfast, NI, United Kingdom

IPD SHARING:
Plan to Share IPD: No